CLINICAL TRIAL: NCT06059859
Title: A Phase III Prospective Randomized Trial to Evaluate the Impact of Augmented Reality During Robot-assisted Radical Prostatectomy on the Rates of Postoperative Surgical Margins
Brief Title: Impact of Augmented Reality During Robot-assisted Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IEO 1310
Record Dates: First submitted 2023-09-13; First posted 2023-09-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented reality robot-assited radical prostatectomy (Experimental): Robot-assisted radical prostatectomy using the Da Vinci surgical robot system (XI model; Intuitive Surgical, Sunnyvale, Calif) and a port device (Alexis; Applied Medical, Rancho Santa Margarita, Calif) system for prostate extraction. Virtual image of the prostate will be overlapped onto the endoscopic view of the Da Vinci surgical robot system using the TilePro system.
  Interventions: Procedure: Augmented reality robot-assited radical prostatectomy; Device: Mixed reality intraoperative frozen section analysis
- Robot-assited radical prostatectomy (Active Comparator): Robot-assisted radical prostatectomy using the Da Vinci surgical robot system (XI model; Intuitive Surgical, Sunnyvale, Calif) and a port device (Alexis; Applied Medical, Rancho Santa Margarita, Calif) system for prostate extraction
  Interventions: Procedure: Robot-assited radical prostatectomy

INTERVENTIONS:
Procedure: Augmented reality robot-assited radical prostatectomy — Robot assisted radical prostatectomy using the Da Vinci surgical robot system (XI model; Intuitive Surgical, Sunnyvale, Calif) and a port device (Alexis; Applied Medical, Rancho Santa Margarita, Calif) system for prostate extraction. Virtual image of the prostate will be overlapped onto the endoscopic view of the Da Vinci surgical robot system using the TilePro system.
  Arms: Augmented reality robot-assited radical prostatectomy
Device: Mixed reality intraoperative frozen section analysis — Microsoft Hololens head-mounted display system will be used for inking prostate margins during intraoperative frozen section analysis
  Arms: Augmented reality robot-assited radical prostatectomy
Procedure: Robot-assited radical prostatectomy — Robot assisted radical prostatectomy using the Da Vinci surgical robot system (XI model; Intuitive Surgical, Sunnyvale, Calif) and a port device (Alexis; Applied Medical, Rancho Santa Margarita, Calif) system for prostate extraction.
  Arms: Robot-assited radical prostatectomy

SUMMARY:
Accurate preservation of neuro-vascular bundles is crucial in guaranteeing erectile function recovery after robot assisted radical prostatectomy (RARP). However, the nerve sparing approach is associated with higher rates of positive surgical margins (PSM) at final pathology. Augmented reality (AR) RARP was previously associated with a 10-15% reduction in the rates of PSMs in two retrospective series. However, prospective studies are needed to demonstrate clinical utility and to validate these technologies. The hypotheses of this study are that: 1) AR RARP reduces the rates of PSMs, if compared to standard approach; 2) AR RARP can guarantee a more accurate preservation of neurovascular bundles and, in consequence, a greater recovery of erectile function; 3) the lower rates of PSMs will translate in greater oncological control of the disease.

DETAILED DESCRIPTION:
This is a Phase III, monocentric, prospective trial in which patients will be randomized to AR RARP vs. standard approach (standard RARP). Patient population is defined as: patients≥18 years old, untreated biopsy-proven adenocarcinoma of the prostate classified as European Association of Urology (EAU) low or intermediate risk (PSA≤20 ng/ml and cT≤2b and International Society for Urological Pathology [ISUP] grade group≤III), pre-operative International Index of Erectile Function-5 (IIEF-5)≥20, no contraindications for multiparametric magnetic resonance imaging (mpMRI). The primary objective of this study is to compare the rates of PSMs with AR RARP vs. standard RARP. Secondary objectives are the rates of nerve sparing approaches and erectile function recovery at 3-, 6- and 12-months after surgery in AR RARP vs. standard RARP. Subgroup analyses will tested for a specific subgroup of patients in which AR RARP should be particularly indicated. Longer-term follow-up will also assess the percentages of biochemical recurrences (BCR) in the two groups.

ELIGIBILITY:
Inclusion Criteria:

Untreated, biopsy-proven adenocarcinoma of the prostate Age ≥18 years

European Association of Urology (EAU) low or intermediate risk prostate cancer:

* PSA≤20 ng/ml
* cT≤2b
* International Society for Urological Pathology [ISUP] grade group≤III Written informed consent provided for participation in the trial International Index of Erectile Function-5 (IIEF-5)≥20 No contraindications for multiparametric magnetic resonance imaging (mpMRI)

Exclusion Criteria:

Any prior therapy for prostate cancer

European Association of Urology (EAU) high risk prostate cancer:

* PSA>20 ng/ml or
* cT>2b or
* ISUP grade group>III International Index of Erectile Function-5 (IIEF-5)<20 Prostate cancer with sarcomatoid or spindle cell or neuroendocrine small cell components Morbidity that would limit compliance with study protocols Controindications to perform mpMRI

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer
Enrollment: 318 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Positive surgical margins | Time zero
  Pathological examination of positive surgical margins according to the criteria of the prostate consensus working group

SECONDARY OUTCOMES:
Surgical time | Time zero
  Total operative time (mins) will we measured from skin incision to skin closure
Nerve-sparing approach | Time zero
  Rates of nerve-sparing approaches between groups will be evaluated according to the Tewari et al. scale
Erectile function | 3-6-12 months after surgery
  Erectile function recovery will be measured with the International Index of Erectile Function-5 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ottavio de Cobelli, MD; PhD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy